CLINICAL TRIAL: NCT01448369
Title: Eyelid Warming Technology for Relief of Meibomian Gland Dysfunction in an Asian Population
Brief Title: Eyelid Warming Technology for Meibomian Gland Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore National Eye Centre (Other Government)
Collaborators: Singapore Eye Research Institute (Other); National University of Singapore (Other)
Responsible Party: Principal Investigator, Louis Tong, Clinician-Scientist, Consultant, Singapore National Eye Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R815/10/2011; 2011/197/A (Other: Singhealth Centralised Institutional Review Board)
Record Dates: First submitted 2011-10-04; First posted 2011-10-07 (Estimated); Last update posted 2014-06-10 (Estimated); Status verified 2014-06

CONDITIONS: Meibomian Gland Dysfunction
Keywords: meibomian gland dysfunction; hot compress; eyelid warming; meibum
MeSH Terms: conditions — Meibomian Gland Dysfunction

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- EyeGiene (Active Comparator): EyeGiene (Eyedetec Medical Inc., US) is a self-contained, convenient warm compress system for the eyes. The system is composed of a reusable eye mask and one time use warmers that are inserted into the eye mask. The warming units are activated by squeezing just prior use and deliver 40°C heat for up to 5 minutes within 30-60 seconds.
  Interventions: Device: EyeGiene
- Blephasteam (Active Comparator): Blephasteam (Spectrum Théa, France) is an eyelid warming device that can be conveniently used at home. The goggles provide standardised heat of about 38 degrees to liquefy lipids and also humidify the chambers with mineral water to ensure optimal moisture levels.
  Interventions: Device: Blephasteam
- Control- Hot Compress (Placebo Comparator): The participants in this group will be using warm compresses with a hot towel.
  Interventions: Device: Hot compresses

INTERVENTIONS:
Device: Blephasteam — 10 minute treatment twice daily
  Other Names: Spectrum Théa, France
  Arms: Blephasteam
Device: EyeGiene — 10 minute treatment, twice daily
  Other Names: Eyedetec Medical Inc., US
  Arms: EyeGiene
Device: Hot compresses — 10 minute treatment, twice daily
  Arms: Control- Hot Compress

SUMMARY:
Meibomian gland dysfunction (MGD), an extremely common clinical condition (seen in more than half of some Asian populations), affects the lipid producing meibomian glands in the eyelids. One function of the glandular secretions is to reduce evaporation of the tear film. In MGD the meibomian glands may become blocked for various reasons. The consequential retention and stasis of the secretion increases immune response as well as scarring response. This eventually results in an abnormal tear film and dry eye symptoms.

The current standard treatments include warm moist compresses, regular lid hygiene, oral antibiotics, topical antibiotic ointments and Omega 3 supplementation. Heating for an extended duration is important because it relieves the occlusion of blocked meibomian glands. However, improvised methods of heating are cumbersome and inefficient requiring repeated measures, often leading to lack of compliance. Today, there is a wider range of commercially available devices that help to unblock meibomian glands and relief dry eye symptoms. These devices may improve MGD treatment dramatically, but have not been tested in the warm climate of Singapore, and are not readily available.

The current study aims to test the efficacy of treatment for devices that utilize A) warm moisture (Blephasteam) and B) warmth (EyeGiene) in patients suffering from meibomian gland dysfunction. Patients will be asked to use Blephasteam and EyeGiene for a period of 4 weeks. The study will monitor patients for changes in tear film and lipid composition, as well as changes in the anatomy of meibomian glands. Additionally, dry eye symptoms will be documented in form of questionnaires. If the newer methods of managing MGD are found to be efficacious and safe, these treatment measures can be made available to patients in Singapore.

DETAILED DESCRIPTION:
Study Objectives and Purpose:

1. A primary purpose of the study is to compare the efficacy of novel eyelid warming devices (Blephasteam and EyeGiene) for treatment of meibomian gland dysfunction by objective clinical scoring and objective assessment of ocular surface parameters in an Asian population.
2. The second aim is to assess the patient acceptance of these modalities, in terms of comfort and convenience.
3. A third aim of the study is to document Meibomian gland disease using non-invasive Meibography, and the possible alterations of this condition after treatment.

Study Design: Prospective, controlled, single masked, interventional study

Rationale:

Meibomian gland dysfunction and resulting evaporative dry eye is highly common in our general population. Behavioral factors and environmental stress may contribute to the severity of the disease. Eyelid warming devices have the potential to significantly improve meibomian gland health and alleviate dry eye symptoms associated with the disease. Currently eyelid warming devices suitable for treatment of meibomian gland dysfunction are not available in Singapore.

Recent technological advances, as well as the infrastructure of the Singapore Eye Research Institute (proximity to Singapore National Eye Center and pre-existing facility and infrastructure for clinical trials) have facilitated studies of products that are available elsewhere and may benefit the Singaporean population.

Methods:

Participants and target sample size Seventy-five patients from the dry eye clinic in the Singapore National Eye Center who have obstructive meibomian gland dysfunction and are keen to test alternative ways for treating the disease will be selected.

Randomisation is done by randomisation table as deemed appropriate by the statistician collaborator.

Treatment regime After informed written consent, patients will be randomly assigned to a group.

1. Control group, 10-minute treatment, twice daily
2. Blephasteam, 10-minute treatment, twice daily
3. EyeGiene, 10-minute treatment, twice daily

All patients are permitted to continue their regular management of MGD such as use of lid scrubs or lid hygiene preparations (such as Lidcare and Blephagel). For consistency, the investigators will monitor the use of such measures in a daily diary and prohibit any other types of treatment for MGD such as Omega-3 tablets, antibiotic or steroid ointments, probing of MG.

Visit schedules Screening visit will be performed at the regular dry eye clinic. If eligible, patients will sign consent and undergo baseline examination.

Subsequent to this, the follow up visit will be after 4 weeks of treatment. A window period of

+/-3days is permitted for this visit.

Duration of study:

Four weeks.

ELIGIBILITY:
Inclusion Criteria:

* Eyelids must present with blocked meibomian gland openings (plugs), at least 1 visible MG plug in the 4 eyelids, or discernable change in consistency of meibum when MG expressed in upper or lower eyelids.
* At least one out of 8 questions on dry eye symptoms is answered with often or all the time (Appendix C, Questionnaire modified after Schein et al.,1997).
* Eyes should not show any other ocular surface pathology which required more treatment than eye lubricant and conventional eyelid hygiene.

Exclusion Criteria:

* Known history of thyroid disorders (diagnosed by physician).
* No ocular surgery within the previous 6 months and LASIK within the previous 1 year.
* Any intake of central nervous system and hormonal drugs within last 30 days and inability to withhold such drugs for at least 6 weeks.
* Active ocular infection or pterygium.
* Anticipated necessity to wear contact lens in the duration of the study.
* Living in the same household as another participant of the study.
* Any other specified reason as determined by clinical investigator, for example, the need to use any treatment or eyedrops (eg. Restasis) not permitted by the study.

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2011-12; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Dry Eye Symptoms | Week 4
  A VAS will be applied to evaluate dry eye symptoms as described by Schaumberg et al. (Schaumberg 2007)between baseline and week 4. The scores will be recorded separately for frequency and severity of dry eye symptoms.

SECONDARY OUTCOMES:
Tear film break up time | Week 4
  After instillation of fluorescein, the participant will be asked to open the eyes, look ahead at the observer's forehead and not blink for as long as possible. The break up time is defined as the time between the lid opening and the first appearance of any dry spot on the cornea. The participant will be requested to close his eyes for few seconds and the procedure will be repeated for the left eye. The tear film break up time will be compared between baseline and week 4.
Number of plugs | Week 4
  The number of blocked/plugged meibomian glands will be counted in each eyelid and any improvement in comparison to baseline assessed.
Yamaguchi Score | Week 4
  The severity of meibomian gland dysfunction will be assessed at baseline and week 4.
Corneal Staining | Week 4
  The corneal staining will be assessed using fluorescein. The cornea will be divided into 5 sectors. The staining will be assessed at baseline and week 4.
Schirmer's Test | Week 4
  The tear production will be assessed using Schirmer Test I. Improvements in tear production will be identified in comparison to baseline.
Meibography | Week 4
  The meibomian glands will be imaged using infrared photography and their health graded at baseline and week 4.
Tear meniscus volume | Week 4
  The tear meniscus (height of the tear film) will be imaged and measured using the Anterior segment optical coherence tomography (AS-OCT). Briefly, the participant will be asked to look at a target in the instrument while blinking normally. The OCT will then scan the ocular surface and images of the upper and lower tear meniscus will be captured. Any changes in tear volume will be assessed with comparison to baseline values.
Meibomian gland lipids | Week 4
  The meibum from patients will be collected using a Kimura Platinum spatula and the lipid components will be analysed using mass-spectrometry. Lipid compositions will be compared between baseline and week 4 visits.
Tear composition | Week 4
  The Schirmer test strips will be collected and the tears analysed for protein and lipid changes at baseline and after 4 weeks of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Louis Tong, PhD, Principal Investigator — Singapore National Eye Centre
Locations (1):
- Singapore National Eye Centre/ Singapore Eye Research Institute, Singapore, Singapore, Singapore

REFERENCES:
- [Background] Lin PY, Tsai SY, Cheng CY, Liu JH, Chou P, Hsu WM. Prevalence of dry eye among an elderly Chinese population in Taiwan: the Shihpai Eye Study. Ophthalmology. 2003 Jun;110(6):1096-101. doi: 10.1016/S0161-6420(03)00262-8. PMID 12799232
- [Background] Foulks GN, Borchman D. Meibomian gland dysfunction: the past, present, and future. Eye Contact Lens. 2010 Sep;36(5):249-53. doi: 10.1097/ICL.0b013e3181ef0d37. PMID 20724853
- [Derived] Yeo S, Tan JH, Acharya UR, Sudarshan VK, Tong L. Longitudinal Changes in Tear Evaporation Rates After Eyelid Warming Therapies in Meibomian Gland Dysfunction. Invest Ophthalmol Vis Sci. 2016 Apr 1;57(4):1974-81. doi: 10.1167/iovs.16-19088. PMID 27096755